CLINICAL TRIAL: NCT03303937
Title: Characteristics of Lower Respiratory Tract Escherichia Coli Isolates Colonizing and Infecting Mechanically Ventilated Intensive Care Patients: a French Multicenter Prospective Collection
Brief Title: Characteristics of Lower Respiratory Tract Escherichia Coli Isolates in Mechanically Ventilated Intensive Care Patients
Acronym: COLOCOLI
Status: Completed | Type: Observational
Sponsor: Hôpital Louis Mourier (Other)
Responsible Party: Principal Investigator, Prof Jean-Damien RICARD, Professor of Intensive Care, Hôpital Louis Mourier
Other Study IDs: HLM_JDR8
Record Dates: First submitted 2017-09-25; First posted 2017-10-06 (Actual); Last update posted 2017-10-06 (Actual); Status verified 2017-10

CONDITIONS: Nosocomial Pneumonia; Ventilator Associated Pneumonia; Escherichia Coli Infections; Escherichia Coli Pneumonia; Escherichia Coli; Diarrhea, Enteroaggregative; Mechanical Ventilation Complication
Keywords: virulence factor genes;; phenotyping; genotyping; antimicrobial susceptibility
MeSH Terms: conditions — Healthcare-Associated Pneumonia; Pneumonia, Ventilator-Associated; Escherichia coli Infections; Diarrhea

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Prospective, multicenter observational study to collect Escherichia coli (E. coli) isolates originating from mechanically ventilated intensive care unit (ICU) patients; in order to characterize phenotype and genotype of E. coli strains retrieved from the lower respiratory tract of ventilated patients.

DETAILED DESCRIPTION:
Prospective, observational, multiple center study performed in 14 ICUs in France to collect Escherichia coli (E. coli) isolates originating from mechanically ventilated intensive care unit (ICU) patients; in order to characterize phenotype and genotype of E. coli strains retrieved from the lower respiratory tract of ventilated patients. All E. coli isolates identified in the microbiology lab and retrieved from a lung specimen (either tracheal aspirate, bronchoalveolar lavage, or telescopic plugged catheter) originating from an ICU patient will be kept, and stored at -80°C in brain-heart infusion broth containing glycerol 20 %. They will be then centralized in the investigators' research unit for further analysis that includes determination of Antimicrobial susceptibility, E. coli phylotype , O-type, and virulence factor gene content.

These isolates will be compared to those of two previously published collections, one from the stools of community subjects, considered as commensal strains, the other from the blood of bacteraemia patients.

ELIGIBILITY:
Inclusion Criteria:

* adult, admitted to the intensive care unit
* under invasive mechanical ventilation
* presence of Escherichia coli in lower respiratory tract specimen

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: any adult critically ill patient admitted to the ICU under invasive mechanical ventilation with a positive lower respiratory tract sample for Escherichia coli
Sampling Method: Probability Sample
Enrollment: 289 (Actual)
Dates: Start 2012-03-27 (Actual); Primary Completion 2015-06-10 (Actual); Study Completion 2016-06-06 (Actual)

PRIMARY OUTCOMES:
phylogenetic group determination | 50 minutes
  Quadruplex polymerase chain reaction (PCR) method was used to determine the E. coli phylogenetic group (A, B1, B2, C, D, E, F), or Escherichia clade I belonging

SECONDARY OUTCOMES:
O-type determination | 50 minutes
  polymerase chain reaction (PCR) method was used to search for the most anticipated serotypes in extra-intestinal infections : O1, O2a, O2b, O4, O6, O7, O12, O15, O16, O17, O18, O22, O25a, O25b, O45a, O75, O78
virulence factor (VF) gene content determination | 90 minutes
  Multiplex PCR was used to detect genes encoding for eleven frequently encountered extraintestinal VFs (S and F fimbriae (sfa/foc), pili associated with pyelonephritis (papC), P adhesin (papGII, papGIII), the ferric yersiniabactin uptake receptor (fyuA), iron transport (iroN), aerobactin (aer), conjugal transfer protein (traT), N-acetylglucosamine 2-epimerase protein (neuC), hemolysin (hlyC), and the cytotoxic necrotizing factor 1(cnf1)
antimicrobial susceptibility determination | 24 hours
  Antimicrobial susceptibility of each isolate was determined by disk-diffusion method according to the French Society of Microbiology. Resistance score was defined as the sum of inactive in vitro antimicrobial agents for each isolate
presence of betalactamase | 90 minutes
  Detection of gene sequences coding for the CTX-M and TEM enzymes was performed by PCR with genomic DNA

OTHER OUTCOMES:
phylogenetic group belonging in other existing Escherichia coli collections | 24 hours
  comparison of phylogenetic group belonging of the present isolates to those of two previously published collections, originating from the Paris area, France; one that comprises 280 E. coli strains isolated from the stools of community adult subjects in 2010 ("COLIVILLE") and that can be considered as commensal strains and the other that comprises 373 E. coli strains isolated from the blood of 373 patients hospitalized in seven different hospitals, during the course of bacteraemia in 2005 (COLIBAFI study)
O-type distribution in other existing Escherichia coli collections | 24 hours
  comparison of O-type distribution of the present isolates to those of two previously published collections, originating from the Paris area, France; one that comprises 280 E. coli strains isolated from the stools of community adult subjects in 2010 ("COLIVILLE") and that can be considered as commensal strains and the other that comprises 373 E. coli strains isolated from the blood of 373 patients hospitalized in seven different hospitals, during the course of bacteraemia in 2005 (COLIBAFI study)
virulence factor (VF) gene content in other existing Escherichia coli collections | 24 hours
  comparison of virulence factor (VF) gene content of the present isolates to those of two previously published collections, originating from the Paris area, France; one that comprises 280 E. coli strains isolated from the stools of community adult subjects in 2010 ("COLIVILLE") and that can be considered as commensal strains and the other that comprises 373 E. coli strains isolated from the blood of 373 patients hospitalized in seven different hospitals, during the course of bacteraemia in 2005 (COLIBAFI study)
phylogenetic group belonging in E. coli isolates responsible for pneumonia and in those responsible for simple colonization | median time frame is 11.5 days with a maximum of 35 days
  comparison of phylogenetic group belonging between isolates responsible for pneumonia and those for simple colonization
O-type distribution in E. coli isolates responsible for pneumonia and in those responsible for simple colonization | median time frame is 11.5 days with a maximum of 35 days
  comparison of O-type distribution between isolates responsible for pneumonia and those for simple colonization
virulence factor (VF) gene content in E. coli isolates responsible for pneumonia and in those responsible for simple colonization | median time frame is 11.5 days with a maximum of 35 days
  comparison of virulence factor (VF) gene content between isolates responsible for pneumonia and those for simple colonization

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Damien Ricard, MD, PhD, Study Director — Assistance Publique - Hôpitaux de Paris; Béatrice La Combe, MD, Principal Investigator — Assistance Publique - Hôpitaux de Paris

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Messika J, Magdoud F, Clermont O, Margetis D, Gaudry S, Roux D, Branger C, Dreyfuss D, Denamur E, Ricard JD. Pathophysiology of Escherichia coli ventilator-associated pneumonia: implication of highly virulent extraintestinal pathogenic strains. Intensive Care Med. 2012 Dec;38(12):2007-16. doi: 10.1007/s00134-012-2699-5. Epub 2012 Sep 28. PMID 23052953
- [Background] Dufour N, Clermont O, La Combe B, Messika J, Dion S, Khanna V, Denamur E, Ricard JD, Debarbieux L; ColoColi group. Bacteriophage LM33_P1, a fast-acting weapon against the pandemic ST131-O25b:H4 Escherichia coli clonal complex. J Antimicrob Chemother. 2016 Nov;71(11):3072-3080. doi: 10.1093/jac/dkw253. Epub 2016 Jul 7. PMID 27387322
- [Background] Massot M, Daubie AS, Clermont O, Jaureguy F, Couffignal C, Dahbi G, Mora A, Blanco J, Branger C, Mentre F, Eddi A, Picard B, Denamur E, The Coliville Group. Phylogenetic, virulence and antibiotic resistance characteristics of commensal strain populations of Escherichia coli from community subjects in the Paris area in 2010 and evolution over 30 years. Microbiology (Reading). 2016 Apr;162(4):642-650. doi: 10.1099/mic.0.000242. Epub 2016 Jan 28. PMID 26822436
- [Background] Lefort A, Panhard X, Clermont O, Woerther PL, Branger C, Mentre F, Fantin B, Wolff M, Denamur E; COLIBAFI Group. Host factors and portal of entry outweigh bacterial determinants to predict the severity of Escherichia coli bacteremia. J Clin Microbiol. 2011 Mar;49(3):777-83. doi: 10.1128/JCM.01902-10. Epub 2010 Dec 22. PMID 21177892
- [Derived] Royer G, Poirel L, La Combe B, Clermont O, Chau F, Mercier-Darty M, Denamur E, Nordmann P, Ricard JD, Decousser JW. Lack of association between colistin resistance and chlorhexidine reduced susceptibility in clinical isolates of Escherichia coli. J Antimicrob Chemother. 2021 Sep 15;76(10):2736-2737. doi: 10.1093/jac/dkab235. No abstract available. PMID 34245272